CLINICAL TRIAL: NCT07251868
Title: Evaluation of Efficacy and Safety of Trop-2 ADC in Breast Cancer Patients With Brain Metastases: A Multicenter Real-World Study
Brief Title: Evaluation of Trop-2 ADC in Breast Cancer Patients With Brain Metastases: A Real-World Study
Status: Recruiting | Type: Observational
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Guohong Song, Chief Physician, Deputy Director of the Department, Medical Oncology of Breast Cancer, Peking University Cancer Hospital & Institute
Other Study IDs: SG-BM-RWS
Record Dates: First submitted 2025-09-24; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer; Brain Metastases From Breast Cancer; Trop2
Keywords: breast cancer; Brain metastases; Trop2; sacituzumab govitecan
MeSH Terms: conditions — Breast Neoplasms; Brain Neoplasms | interventions — sacituzumab govitecan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients received Trop-2 ADC （SG）: Advanced breast cancer patients with brain metastases who were treated with Sacituzumab Govitecan (SG).
  Interventions: Drug: Sacituzumab Govitecan (SG)

INTERVENTIONS:
Drug: Sacituzumab Govitecan (SG) — Sacituzumab Govitecan
  Other Names: IMMU-132; Sacituzumab Govitecan-hziy

SUMMARY:
The goal of this real-world study (RWS) is to evaluate the effectiveness of Trop-2 ADC (sacituzumab govitecan) in treating breast cancer patients with brain metastases, and to understand the safety profile of this drug in real clinical practice across multiple centers. The main questions it aims to answer are:

Does Trop-2 ADC (sacituzumab govitecan) improve intracranial outcomes in breast cancer patients with brain metastases (e.g., intracranial objective response rate, intracranial progression-free survival)? What types and rates of adverse events do breast cancer patients with brain metastases experience when receiving Trop-2 ADC (sacituzumab govitecan)? This is a multicenter real-world study, which will collect and analyze data from breast cancer patients with brain metastases who have received Trop-2 ADC (sacituzumab govitecan) in routine clinical care (no randomization or placebo control, consistent with real-world clinical scenarios).

Participants (breast cancer patients with brain metastases who received Trop-2 ADC) will have their data collected from:

Electronic health records (EHRs) across multiple medical centers Regular clinical follow-up visits (e.g., once every 4-8 weeks) for imaging assessments (to evaluate brain metastasis changes) and safety monitoring Medical records documenting treatment responses, disease progression, and any adverse events during treatment and follow-up

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old (based on actual age at the time of signing the informed consent form), with no restriction on gender
* Able to understand the study purpose, risks, and benefits, and voluntarily sign the written informed consent form; if the patient has cognitive impairment or is unable to express themselves independently, their legal guardian/authorized agent shall sign after being fully informed, and provide valid authorization documents.
* Have access to complete medical records (including breast cancer primary lesion diagnosis data, brain metastasis diagnosis data, SG treatment records, follow-up data, etc.) in the study collaborating medical institutions/specified medical systems to ensure traceability of treatment processes and outcomes.

Diagnosed with breast cancer via histopathological/cytopathological examination, with the diagnostic report issued by a tertiary hospital or the study-designated pathology center.

* Diagnosed with breast cancer brain metastasis based on meeting any of the following conditions: ① Definitive diagnosis by a physician with associate senior title or above, combining contrast-enhanced cranial magnetic resonance imaging (MRI)/computed tomography (CT) with clinical symptoms and signs; ② Postoperative pathology of brain metastatic lesions confirming breast cancer metastasis; ③ Pathological examination of brain metastatic lesion biopsy specimens confirming breast cancer metastasis.
* No restrictions on the number, size of brain metastatic lesions, presence of meningeal metastasis, or presence of brain metastasis-related symptoms (e.g., headache, limb dysfunction).
* Previous treatment with Sacituzumab Govitecan (SG), with clear medication records (prescription orders, medical orders, pharmacy dispensing records, etc.), and no restrictions on the line of SG treatment, dosage, or treatment cycles (both completion of full-cycle treatment and early discontinuation due to adverse reactions/progression are acceptable).
* No restriction on the start time of SG treatment ; patients currently receiving SG treatment, who have completed SG treatment, or who have discontinued SG treatment due to objective reasons are all eligible.
* Stable vital signs at present, without the following uncontrolled severe conditions: ① Severe infections such as sepsis and severe pneumonia (symptoms relieved and laboratory indicators normalized after anti-infective treatment); ② Epileptic seizures within the past 3 months (or uncontrolled without standardized anti-epileptic treatment); ③ Failure of major organs such as heart, liver, and kidney (e.g., New York Heart Association (NYHA) Class Ⅳ cardiac function, Child-Pugh Class C liver function, chronic kidney disease Stage 5) .
* The patient/guardian can cooperate with study follow-up (outpatient follow-up, telephone follow-up, electronic medical record extraction, etc.), and survival status, disease progression, subsequent treatment, adverse reactions, and other information can be obtained within the expected follow-up period.

Exclusion Criteria:

* Complicated with other primary malignant tumors (excluding breast cancer), and the tumor was in an active stage within the past 5 years (not achieving complete remission or disease-free survival for more than 5 years).
* Unable to cooperate with informed consent or follow-up due to mental illness, cognitive impairment, etc., and without qualified guardian assistance.
* Concurrent participation in other interventional clinical trials (e.g., randomized controlled trials), which may affect data collection and result interpretation of this study.
* Other conditions judged by the researcher to affect study quality or patient safety .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with breast cancer and brain metastases, aged ≥18 years, who have received Sacituzumab Govitecan (SG).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Real world progression free survival (rwPFS) | up to 48 months from the initiation of the study treatment.
  The time interval from the date of Sacituzumab Govitecan initiation until date of progressive disease (PD) or death from any causes, whichever occurred first.

SECONDARY OUTCOMES:
Real world objective response rate (rwORR) | approximately up to 24 weeks from the initiation of the study treatment.
  The percentage of participants with the best overall response of complete response (CR) or partial response (PR) according to RECIST 1.1. CR = Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR = At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Real world overall survival (rwOS) | up to 48 months from the initiation of the study treatment.
  Time from initiation of SG monotherapy or combination therapy to death from any cause
Number of patients with adverse events | approximately up to 68 weeks from the initiation of the treatment.
  Adverse events were assessed during study treatment and at follow-up visits
CNS-PFS | Start of treatment until 2-year follow-up
  Central nervous system- progression free survival: time from the date when the subject first received SG to the first observation of tumor progression of central nervous system or death from any cause.
CNS-ORR | Start of treatment until 2-year follow-up
  Central nervous system- objective response rate: proportion of subjects who achieved complete remission (CR) or partial remission (PR) of central nervous system by primary tumor imaging evaluation.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided